CLINICAL TRIAL: NCT01725451
Title: Effects of Deodorant and Antiperspirant Use and the Presence of Axillary Hair on the Absorption of Testosterone Applied as Testosterone 2% Solution
Brief Title: A Study of Effect of Deodorant and Axillary Hair on Testosterone Absorption in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15083; I5E-MC-TSBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Testosterone; Testosterone Propionate; Deodorants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Testosterone Unshaved (Experimental): No deodorant or antiperspirant: Single 30 mg dose of testosterone applied topically to each unshaved axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone
- Testosterone Unshaved + Deodorant Spray (Experimental): Deodorant spray applied to unshaved axillae. At least 2 minutes wait time. Then, single 30 mg dose of testosterone applied topically to each axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone; Other: Deodorant Spray
- Testosterone Unshaved + Deodorant Antiperspirant Spray (Experimental): Deodorant antiperspirant combination spray applied to unshaved axillae. At least 2 minutes wait time. Then, single 30 mg dose of testosterone applied topically to each axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone; Other: Deodorant and Antiperspirant Combination Spray
- Testosterone Unshaved + Deodorant Antiperspirant Stick (Experimental): Deodorant antiperspirant combination stick applied to unshaved axillae. At least 2 minutes wait time. Then, single 30 mg dose of testosterone applied topically to each axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone; Other: Deodorant and Antiperspirant Combination Stick
- Testosterone Shaved (Experimental): No deodorant or antiperspirant: Single 30 mg dose of testosterone applied topically to each shaved axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone
- Testosterone Shaved + Deodorant Antiperspirant Spray (Experimental): Deodorant antiperspirant combination spray applied to shaved axillae. At least 2 minutes wait time. Then, single 30 mg dose of testosterone applied topically to each axilla in 1 of 6 treatment periods.
  Interventions: Drug: Testosterone; Other: Deodorant and Antiperspirant Combination Spray

INTERVENTIONS:
Drug: Testosterone — Administered topically to axillae
  Other Names: Axiron; LY900011
Other: Deodorant Spray — Administered topically to axillae
  Arms: Testosterone Unshaved + Deodorant Spray
Other: Deodorant and Antiperspirant Combination Spray — Administered topically to axillae
  Arms: Testosterone Shaved + Deodorant Antiperspirant Spray; Testosterone Unshaved + Deodorant Antiperspirant Spray
Other: Deodorant and Antiperspirant Combination Stick — Administered topically to axillae
  Arms: Testosterone Unshaved + Deodorant Antiperspirant Stick

SUMMARY:
This study will evaluate the effect of deodorant and antiperspirant use and the presence of underarm hair on the absorption of testosterone. Each participant in this study will receive 6 single doses of 30 milligrams (mg) testosterone applied as a solution to each underarm. There is a minimum one day washout period between each dose. This study will last approximately 24 days not including screening. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males, as determined by medical history and physical examination
* Agree to use a reliable method of birth control (for example, condom or vasectomy) during the study and for 1 month following the last dose of testosterone
* Have a total testosterone level <400 nanograms per deciliter (ng/dL) based on local laboratory result
* Have a hemoglobin ≥12 grams per deciliter (g/dL) at screening and, if the participant takes a break from the study, at the re-test
* Weigh at least 60 kilograms (kg)
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Eli Lilly and Company (Lilly) and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Use any topical testosterone replacement therapy within the 2 weeks prior to randomization through the last dosing period, except for use of testosterone solution as directed by study procedures
* Use parenteral testosterone replacement (testosterone enanthanate, testosterone cypionate) within the 30 days prior to screening. Use long-acting intramuscular testosterone undecanoate 6 months prior to screening, or use of testosterone pellets 12 months prior to screening
* Have a body mass index >35 kilograms per square meter (kg/m^2)
* Have a significant history of allergy and/or sensitivity to the drug products or excipients, including any history of sensitivity to testosterone
* Currently use any medications, herbal, and/or nutritional supplements that can interfere with testosterone
* Have a dermatologic condition in the underarm area that might interfere with testosterone absorption (for example, eczema) or be exacerbated by topical testosterone replacement therapy
* Have a history or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, endocrine, hematological, or neurological disorders constituting a risk when taking the study medication of that could interfere with the interpretation of the data
* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Have an abnormal prostate-specific antigen (PSA) test result
* Have known allergies to testosterone solution, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure as determined by the investigator
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of human immunodeficiency (HIV) infection and/or positive human HIV antibodies
* Are participants who have previously completed or withdrawn from this study or any other study investigating testosterone
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or nonapproved use of a drug or device (other than the investigational product used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study
* Have shaved the axillae within 3 months of screening

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana

REFERENCES:
- [Derived] Small DS, Ni X, Polzer P, Vart R, Satonin DK, Mitchell MI. Effect of deodorant and antiperspirant use and presence or absence of axillary hair on absorption of testosterone 2% solution applied to men's axillae. J Sex Med. 2014 Nov;11(11):2809-17. doi: 10.1111/jsm.12658. Epub 2014 Aug 14. PMID 25123988

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: 30-milligram (mg) testosterone 2% solution applied to each unshaved axilla without deodorant or antiperspirant in Period 1, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination stick in Period 2, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant spray in Period 3, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination spray in Period 4, 30-mg testosterone 2% solution applied to each shaved axilla without deodorant or antiperspirant in Period 5, and 30-mg testosterone 2% solution applied to each shaved axilla with deodorant/antiperspirant combination spray in Period 6. Each of the treatments was followed by 3 days of pharmacokinetic (PK) sampling and 1-day washout except that there was no washout after the last PK sample for the last treatment.
- Sequence 2: 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant spray in Period 1, 30-mg testosterone 2% solution applied to each unshaved axilla without deodorant or antiperspirant in Period 2, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination spray in Period 3, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination stick in Period 4, 30-mg testosterone 2% solution applied to each shaved axilla with deodorant/antiperspirant combination spray in Period 5, 30-mg testosterone 2% solution applied to each shaved axilla without deodorant or antiperspirant in Period 6. Each of the treatments was followed by 3 days of pharmacokinetic (PK) sampling and 1-day washout except that there was no washout after the last PK sample for the last treatment.
- Sequence 3: 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination spray in Period 1, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant spray in Period 2, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination stick in Period 3, 30-mg testosterone 2% solution applied to each unshaved axilla without deodorant or antiperspirant in Period 4, 30-mg testosterone 2% solution applied to each shaved axilla without deodorant or antiperspirant in Period 5, and 30-mg testosterone 2% solution applied to each shaved axilla with deodorant/antiperspirant combination spray in Period 6. Each of the treatments was followed by 3 days of pharmacokinetic (PK) sampling and 1-day washout except that there was no washout after the last PK sample for the last treatment.
- Sequence 4: 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination stick in Period 1, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant/antiperspirant combination spray in Period 2, 30-mg testosterone 2% solution applied to each unshaved axilla without deodorant or antiperspirant in Period 3, 30-mg testosterone 2% solution applied to each unshaved axilla with deodorant spray in Period 4, 30-mg testosterone 2% solution applied to each shaved axilla with deodorant/antiperspirant combination spray in Period 5, and 30-mg testosterone 2% solution applied to each shaved axilla without deodorant or antiperspirant in Period 6. Each of the treatments was followed by 3 days of pharmacokinetic (PK) sampling and 1-day washout except that there was no washout after the last PK sample for the last treatment.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 7 | 8 | 7
Completed | 7 | 7 | 8 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Washout From Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 7 | 8 | 7
Completed | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 7 | 8 | 7
Completed | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout From Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 7 | 8 | 7
Completed | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 7 | 8 | 7
Completed | 7 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout From Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 7 | 8 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 7 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Washout From Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout From Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 6 | 7
Completed | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of testosterone 2% solution.
Groups:
- Testosterone 2% Solution: Participants randomized to 1 of 4 treatment sequences involving 6 treatments in each sequence. Each sequence involved 4 single-dose treatments of testosterone 2% solution to unshaved axillae with or without the use of deodorant or antiperspirant products followed by 2 single-dose treatments of testosterone 2% solution to shaved axillae with or without the use of deodorant or antiperspirant products. Each of the treatments was followed by 3 days of pharmacokinetic (PK) sampling and 1-day washout except that there was no washout after the last PK sample for the last treatment.
Arm/Group | Testosterone 2% Solution
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native/White | 1
  Black or African American | 1
  White | 28
Region of Enrollment [Number; unit: participants]
  United States | 30
Screening Testosterone [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] | 290.8 (78.2)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of Testosterone
Description: The AUC from time 0 to 72 hours [AUC (0-72)] postdose, based on baseline-corrected concentrations. Baseline-corrected AUC (0-72) was calculated using the measured concentrations of total testosterone minus mean baseline testosterone concentration. Baseline testosterone concentration was the arithmetic mean of 3 predose concentrations.
Time Frame: Pre-dose [60 to 45 minutes (min), 30 to 15 min, 5 minutes prior to each dose], 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, and 72 hours after administration of study drug
Population: All randomized participants who received at least 1 dose of testosterone 2% solution and had evaluable 72-hour testosterone concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms* hours per deciliter (ng*h/dL)
Groups:
- Testosterone Unshaved: No deodorant or antiperspirant. A single 30-milligram (mg) dose of testosterone 2% solution applied topically to each unshaved axilla.
- Testosterone Unshaved + Deodorant Spray: Deodorant spray applied to each unshaved axilla ≥2 minutes before application of a single 30-mg dose of testosterone 2% solution.
- Testosterone Unshaved + Deodorant Antiperspirant Spray: Deodorant antiperspirant combination spray applied to each unshaved axilla ≥2 minutes before application of a single 30-mg dose of testosterone 2% solution.
- Testosterone Unshaved + Deodorant Antiperspirant Stick: Deodorant/antiperspirant combination stick applied to each unshaved axilla ≥2 minutes before application of a single 30-mg dose of testosterone 2% solution.
- Testosterone Shaved: No deodorant or antiperspirant. A single 30-mg dose of testosterone 2% solution applied topically to each shaved axilla.
- Testosterone Shaved + Deodorant Antiperspirant Spray: Deodorant/antiperspirant combination spray applied to each shaved axilla ≥2 minutes before application of a single 30-mg dose of testosterone 2% solution.
Arm/Group | Testosterone Unshaved | Testosterone Unshaved + Deodorant Spray | Testosterone Unshaved + Deodorant Antiperspirant Spray | Testosterone Unshaved + Deodorant Antiperspirant Stick | Testosterone Shaved | Testosterone Shaved + Deodorant Antiperspirant Spray
Number analyzed (Participants) | 27 | 29 | 29 | 28 | 26 | 26
nanograms* hours per deciliter (ng*h/dL) | 2120 (164.0) | 2400 (196.0) | 2970 (92.0) | 2880 (129.0) | 3110 (129.0) | 2070 (1733.0)

2. Primary Outcome: Pharmacokinetics: Maximum Drug Concentration (Cmax) of Testosterone
Description: The Cmax from time 0 to 72 hours postdose, based on baseline-corrected concentrations. Baseline-corrected Cmax was calculated using the measured concentrations of total testosterone minus mean baseline testosterone concentration. Baseline testosterone concentration was the arithmetic mean of 3 predose concentrations.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of testosterone 2% solution for the specified treatment regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per deciliter (ng/dL)
Groups:
- Testosterone Unshaved + Deodorant Antiperspirant Spray: Deodorant antiperspirant combination spray applied to each unshaved axilla ≥2 minutes before application of a single 30-mg dose of testosterone 2% solution .
Arm/Group | Testosterone Unshaved | Testosterone Unshaved + Deodorant Spray | Testosterone Unshaved + Deodorant Antiperspirant Spray | Testosterone Unshaved + Deodorant Antiperspirant Stick | Testosterone Shaved | Testosterone Shaved + Deodorant Antiperspirant Spray
Number analyzed (Participants) | 29 | 29 | 29 | 28 | 26 | 26
nanograms per deciliter (ng/dL) | 214 (97.0) | 209 (119.0) | 234 (106.0) | 202 (97.0) | 231 (102.0) | 151 (519.0)

ADVERSE EVENTS:
Arm/Group | Testosterone Unshaved | Testosterone Unshaved + Deodorant Spray | Testosterone Unshaved + Deodorant Antiperspirant Spray | Testosterone Unshaved + Deodorant Antiperspirant Stick | Testosterone Shaved | Testosterone Shaved + Deodorant Antiperspirant Spray
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/28 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/29 | 1/29 | 2/29 | 4/28 | 0/26 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Unshaved (N=29) | Testosterone Unshaved + Deodorant Spray (N=29) | Testosterone Unshaved + Deodorant Antiperspirant Spray (N=29) | Testosterone Unshaved + Deodorant Antiperspirant Stick (N=28) | Testosterone Shaved (N=26) | Testosterone Shaved + Deodorant Antiperspirant Spray (N=26)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days